CLINICAL TRIAL: NCT07338370
Title: Relation Between Prostaglandin E2 Metabolite Levels and the Development of Hemodynamically Significant Patent Ductus Arteriosus in Preterm Neonates
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD143/2025
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Prematurity; Patent Ductus Arteriosus in Preterm Infants; Prostaglandins
Keywords: cerebral blood flow; neonates; PDA; preterms
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PGE2

GROUPS / COHORTS (2):
- group1, hemodynamically significant PDA: fulfilling the following criteria PDA measuring > 1.5 mm and predominantly left-to-right shunt. LA/Ao ratio between 1.4 and 1.6 in moderate PDA and >1.6 in large PDA. Left pulmonary artery (LPA) diastolic flow velocity of >0.25 m/sec. Systemic hypo perfusion: absent or reversed diastolic flow in the Aorta Group1will receive anti-PGE; Ibuprofen (IBU) (brufen)® syrup will be given for 3 days enterally either orally or via a gastric tube with an initial dose of 10mg/kg/day, followed by 5mg/kg/day for the next 2 days
  Interventions: Drug: Ibuprofen (Brufen®)
- group2, hemodynamically insignificant PDA: Spontaneous closure group by echocardiography

INTERVENTIONS:
Drug: Ibuprofen (Brufen®) — Group1will receive anti-PGE; Ibuprofen (IBU) (brufen)® syrup will be given for 3 days enterally either orally or via a gastric tube with an initial dose of 10mg/kg/day, followed by 5mg/kg/day for the next 2 days.
  Group 2 will be observed and follow up echocardiography and PGE2 level will be followed up 3 days after treatment or follow up in both groups.
  Groups: group1, hemodynamically significant PDA

SUMMARY:
prospective observational cohort study to explore the relationship between PGE2 metabolite levels and the development of hemodynamically significant PDA in preterm neonates.

DETAILED DESCRIPTION:
Regulation of ductus arteriosus involves (PGE2), produced by the placenta and DA itself, that promotes ductal patency by relaxing smooth muscle.

Prostaglandins are pluripotent lipid mediators derived from membrane glycerophospholipid metabolism. They are synthesized via a multienzyme cascade involving the actions of phospholipases and COX isoforms. Prostanoids, such as prostaglandin E2 and prostaglandin D2 metabolite (PGDM), are produced by various structural and inflammatory cells.

Cyclooxygenase inhibitors restrict the PDA by inhibiting the prostaglandin synthase enzyme, which prevents arachidonic acid from converting to prostaglandin. Acetaminophen is also believed to inhibit the prostaglandin synthesis enzyme's peroxidase portion, resulting in the PDA narrowing.

A significant decrease in serum PGE2 levels was observed following COX inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates with gestational age ≤ 32 weeks, admitted to the NICU and diagnosed with patent ductus arteriosus by echocardiography on day 3 of life.

Exclusion Criteria:

* Preterm neonates with evidence of any of the following will be excluded:

Chromosomal anomaly or Congenital malformations Progressive intraventricular hemorrhage Congenital heart defect other than PDA and/or patent foramen ovale Pulmonary hypertension with right to left shunt on PDA Contraindications to the use of Ibuprofen: [1] Urine output <1 mL/kg/hour during preceding 8 hours. Serum creatinine >1.6 mg/dL. Platelet count <50 000/mm3. Abnormal coagulation profile. Necrotizing enterocolitis (NEC) or intestinal perforation

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates admitted to Ain shams University Hospital NICUs fulfilling the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Explore the relationship between PGE2 metabolite levels and the development of hemodynamically significant PDA in preterm neonates. | initial PGE2 level on the first day of life and follow up the level after 3 days of treatment
  correlating the initial levels of PGE2 with the significance of PDA

CONTACTS AND LOCATIONS:
Overall Officials: Mennatallah Ayman ayman, masters, Principal Investigator — Neonatal intensive care units (NICUs), Ain Shams University, Abbasia, Cairo, Egypt, 11517
Locations (1):
- Faculty of Medicine, Ain Shams, University, Cairo, Abbasia, Egypt